CLINICAL TRIAL: NCT03575351
Title: A Global Randomized Multicenter Phase 3 Trial of JCAR017 Compared to Standard of Care in Adult Subjects With High-risk, Second-line, Transplant-eligible Relapsed or Refractory Aggressive B-cell Non-Hodgkin Lymphomas (TRANSFORM).
Brief Title: A Study to Compare the Efficacy and Safety of JCAR017 to Standard of Care in Adult Subjects With High-risk, Transplant-eligible Relapsed or Refractory Aggressive B-cell Non-Hodgkin Lymphomas
Acronym: TRANSFORM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCAR017-BCM-003; U1111-1213-1944 (Registry Identifier: WHO); 2018-000929-32 (EudraCT Number)
Record Dates: First submitted 2018-06-14; First posted 2018-07-02 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Non-Hodgkin Lymphomas; DLBCL; Efficacy; Safety; JCAR017; Liso-cel; High-Risk; Relapsed; Refractory; B-cell NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Standard of Care (SOC) (Active Comparator): Subjects should receive SOC (R-DHAP, R-ICE or R-GDP) followed by HDCT (BEAM) and HSCT. Standard of care regimen will be administered as per investigator decision.
  Interventions: Drug: Standard of Care
- Arm B - JCAR017 (Experimental): Lymphodepleting chemotherapy with intravenous (IV) fludarabine (30 mg/m2/day for 3 days) plus cyclophosphamide IV (300 mg/m2/day for 3 days) (flu/cy) concurrently followed by JCAR017 infusion.
  Interventions: Genetic: JCAR017

INTERVENTIONS:
Drug: Standard of Care — Standard of Care
  Arms: Arm A - Standard of Care (SOC)
Genetic: JCAR017 — JCAR017
  Other Names: lisocabtagene maraleucel or liso-cel
  Arms: Arm B - JCAR017

SUMMARY:
The study will be conducted in compliance with the International Council for Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

This is a randomized, open-label, parallel-group, multi-center trial in adult subjects with Relapsed or refractory (R/R) aggressive Non-Hodgkin lymphoma (NHL) to compare safety and efficacy between the standard of care (SOC) strategy versus JCAR017 (also known as lisocabtagene maraleucel or liso-cel). Subjects will be randomized to either receive SOC (Arm A) or to receive JCAR017 (Arm B).

All subjects randomized to Arm A will receive Standard of care (SOC) salvage therapy (R-DHAP, RICE or R-GDP) as per physician's choice before proceeding to High dose chemotherapy (HDCT) and Hematopoietic stem cell transplant (HSCT).

Subjects from Arm A may be allowed to cross over and receive JCAR017 upon confirmation of an EFS event.

Subjects randomized to Arm B will receive Lymphodepleting (LD) chemotherapy followed by JCAR017 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years and ≤ 75 years of age at the time of signing the informed consent form (ICF).
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
3. Histologically proven diffuse large B-cell lymphoma (DLBCL) NOS (de novo or transformed indolent NHL), high grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements with DLBCL histology (double/triple-hit lymphoma [DHL/THL]), primary mediastinal (thymic) large B-cell lymphoma (PMBCL), T cell/histiocyte-rich large B-cell lymphoma (THRBCL) or follicular lymphoma grade 3B. Enough tumor material must be available for confirmation by central pathology.
4. Refractory or relapsed within 12 months from CD20 antibody and anthracycline containing first line therapy.
5. [18F] fluorodeoxyglucose (FDG) positron emission tomography (PET) positive lesion at screening. (Deauville score 4 or 5)
6. Adequate organ function
7. Participants must agree to use effective contraception

Exclusion Criteria:

1. Subjects not eligible for hematopoietic stem cell transplantation (HSCT).
2. Subjects planned to undergo allogeneic stem cell transplantation.
3. Subjects with, primary cutaneous large B-cell lymphoma, EBV (Epstein-Barr virus) positive DLBCL, Burkitt lymphoma or transformation from chronic lymphocytic leukemia/small lymphocytic lymphoma (Richter transformation).
4. Subjects with prior history of malignancies, other than aggressive R/R NHL, unless the subject has been free of the disease for ≥ 2 years with the exception of the following noninvasive malignancies:

   * Basal cell carcinoma of the skin
   * Squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is curative.
   * Other completely resected stage 1 solid tumor with low risk for recurrence
5. Treatment with any prior gene therapy product.
6. Subjects who have received previous CD19-targeted therapy.
7. Subjects with active hepatitis B, or active hepatitis C are excluded. Subjects with negative polymerase chain reaction (PCR) assay for viral load for hepatitis B or C are permitted. Subjects positive for hepatitis B surface antigen and/or anti-hepatitis B core antibody with negative viral load are eligible and should be considered for prophylactic antiviral therapy. Subjects with a history of or active human immunodeficiency virus (HIV) are excluded.
8. Subjects with uncontrolled systemic fungal, bacterial, viral or other infection (including tuberculosis) despite appropriate antibiotics or other treatment.
9. Active autoimmune disease requiring immunosuppressive therapy.
10. History of any one of the following cardiovascular conditions within the past 6 months prior to signing the ICF: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease.
11. History or presence of clinically relevant central nervous system (CNS) pathology
12. Pregnant or nursing (lactating) women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (54):
- United States (28):
  - Local Institution - 129, Scottsdale, Arizona
  - Local Institution - 116, Scottsdale, Arizona
  - Local Institution - 115, San Francisco, California
  - Local Institution - 106, Aurora, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Local Institution - 126, Tampa, Florida
  - Local Institution - 108, Atlanta, Georgia
  - Local Institution - 107, Atlanta, Georgia
  - Local Institution - 122, Chicago, Illinois
  - Loyola University Medical Center Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Local Institution - 102, Boston, Massachusetts
  - Local Institution - 104, Boston, Massachusetts
  - Local Institution - 120, Ann Arbor, Michigan
  - Local Institution - 119, Detroit, Michigan
  - Local Institution - 112, Minneapolis, Minnesota
  - Local Institution - 103, Rochester, Minnesota
  - Local Institution - 100, Omaha, Nebraska
  - Local Institution - 121, Hackensack, New Jersey
  - Local Institution - 111, Buffalo, New York
  - Local Institution - 117, New York, New York
  - Local Institution - 125, Charlotte, North Carolina
  - Local Institution - 127, Oklahoma City, Oklahoma
  - Local Institution - 101, Portland, Oregon
  - Local Institution - 123, Pittsburgh, Pennsylvania
  - Local Institution - 109, Dallas, Texas
  - Local Institution - 124, Houston, Texas
  - Local Institution - 114, Richmond, Virginia
  - Local Institution - 110, Seattle, Washington
- Local Institution - 350, Ghent, Belgium
- Local Institution - UNK 25, Helsinki, Finland
- France (4):
  - Local Institution - 401, Lille
  - Local Institution - 400, Marseille
  - Local Institution - 403, Pierre-Bénite
  - Local Institution - 402, Villejuif
- Germany (6):
  - Local Institution - 455, Dresden, Saxony
  - Local Institution - 451, Berlin
  - Local Institution - 450, Cologne
  - Local Institution - 452, Hamburg
  - Local Institution - 453, München
  - Local Institution - 454, Münster
- Italy (3):
  - Local Institution - 500, Rome
  - Local Institution - 501, Rozzano (MI)
  - Local Institution - 502, Torino
- Japan (4):
  - Local Institution - 203, Osaka, Osaka-shi
  - Local Institution - 200, Chuo-ku, Tokyo
  - Local Institution - 201, Minato-ku, Tokyo
  - Local Institution - 202, Bunkyō City
- Local Institution - 550, Rotterdam, Netherlands
- Spain (2):
  - Local Institution - 600, Barcelona
  - Local Institution - 601, Madrid
- Local Institution - 650, Stockholm, Sweden
- Local Institution - 700, Bern, Switzerland
- United Kingdom (2):
  - Local Institution - 751, Southampton, Hampshire
  - Local Institution - 750, London

REFERENCES:
- [Derived] Kamdar M, Solomon SR, Arnason J, Johnston PB, Glass B, Bachanova V, Ibrahimi S, Mielke S, Mutsaers P, Hernandez-Ilizaliturri F, Izutsu K, Morschhauser F, Lunning M, Chow VA, Montheard S, Santamaria J, Colicino S, Ogasawara K, Stepan L, Liu FF, Abramson JS. Lisocabtagene Maraleucel Versus Standard of Care for Second-Line Relapsed/Refractory Large B-Cell Lymphoma: 3-Year Follow-Up From the Randomized, Phase III TRANSFORM Study. J Clin Oncol. 2025 Aug 20;43(24):2671-2678. doi: 10.1200/JCO-25-00399. Epub 2025 Jul 7. PMID 40623279
- [Derived] Abramson JS, Solomon SR, Arnason J, Johnston PB, Glass B, Bachanova V, Ibrahimi S, Mielke S, Mutsaers P, Hernandez-Ilizaliturri F, Izutsu K, Morschhauser F, Lunning M, Crotta A, Montheard S, Previtali A, Ogasawara K, Kamdar M. Plain language summary of the TRANSFORM study primary analysis results: liso-cell as a second treatment regimen for large B-cell lymphoma following failure of the first treatment regimen. Future Oncol. 2024;20(21):1455-1465. doi: 10.2217/fon-2023-0898. Epub 2024 Mar 28. PMID 38547003
- [Derived] Saeedian M, Badaracco J, Botros A, Gitlin M, Keating SJ. Estimating the Cost per Clinical Outcome of Second-Line Liso-Cel Versus Autologous Stem Cell Transplantation in Patients with Transplantation-Intended Relapsed/Refractory Large B Cell Lymphoma. Transplant Cell Ther. 2023 Nov;29(11):712.e1-712.e7. doi: 10.1016/j.jtct.2023.08.001. Epub 2023 Aug 5. PMID 37544410
- [Derived] Abramson JS, Solomon SR, Arnason J, Johnston PB, Glass B, Bachanova V, Ibrahimi S, Mielke S, Mutsaers P, Hernandez-Ilizaliturri F, Izutsu K, Morschhauser F, Lunning M, Crotta A, Montheard S, Previtali A, Ogasawara K, Kamdar M. Lisocabtagene maraleucel as second-line therapy for large B-cell lymphoma: primary analysis of the phase 3 TRANSFORM study. Blood. 2023 Apr 6;141(14):1675-1684. doi: 10.1182/blood.2022018730. PMID 36542826
- [Derived] Kamdar M, Solomon SR, Arnason J, Johnston PB, Glass B, Bachanova V, Ibrahimi S, Mielke S, Mutsaers P, Hernandez-Ilizaliturri F, Izutsu K, Morschhauser F, Lunning M, Maloney DG, Crotta A, Montheard S, Previtali A, Stepan L, Ogasawara K, Mack T, Abramson JS; TRANSFORM Investigators. Lisocabtagene maraleucel versus standard of care with salvage chemotherapy followed by autologous stem cell transplantation as second-line treatment in patients with relapsed or refractory large B-cell lymphoma (TRANSFORM): results from an interim analysis of an open-label, randomised, phase 3 trial. Lancet. 2022 Jun 18;399(10343):2294-2308. doi: 10.1016/S0140-6736(22)00662-6. PMID 35717989
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Thiruvengadam SK, Hunter B, Varnavski A, Fakhri B, Kaplan L, Ai WZ, Pampaloni M, Huang CY, Martin T 3rd, Damon L, Andreadis CB. Ofatumumab, Etoposide, and Cytarabine Intensive Mobilization Regimen in Patients with High-risk Relapsed/Refractory Diffuse Large B-Cell Lymphoma Undergoing Autologous Stem Cell Transplantation. Clin Lymphoma Myeloma Leuk. 2021 Apr;21(4):246-256.e2. doi: 10.1016/j.clml.2020.11.005. Epub 2020 Nov 11. PMID 33288485
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care Arm: 3 cycles of standard of care (SOC) salvage therapy (rituximab, dexamethasone, cytarabine and cisplatin [R-DHAP], rituximab, ifosfamide, carboplatin and etoposide [R-ICE], rituximab, gemcitabine, dexamethasone, and cisplatin [R-GDP]) per physician's choice. Participants responding to SOC are expected to undergo high dose chemotherapy (HDCT) and hematopoietic stem cell transplant (HSCT). If requested by the investigator, participants may be allowed to receive JCAR017 upon meeting progression, relapse, or suboptimal response. 1 cycle = 3 weeks
- Liso-cel Arm: [Lymphodepleting chemotherapy (LDC)] Fludarabine IV (30 mg/m^2/day for 3 days) and cyclophosphamide IV (300 mg/m^2/day for 3 days) followed by JCAR017 IV infusion at a dose of 100 x 10^6 JCAR017-positive viable transduced T cells (CAR+ T cells) on Day 29 (2 to 7 days after completion of LD chemotherapy)
Period: Overall Study
Arm/Group | Standard of Care Arm | Liso-cel Arm
Started (Randomized) | 92 | 92 (Received lymphodepleting chemotherapy (LDC))
Treated | 91 (SOC Treatment) | 90 (Liso-cel Treatment)
Crossover (Received SOC but were eligible to receive JCAR017 treatment) | 61 | 0
Received JCAR017 Conforming Cell Product | 57 | 89
Received JCAR017 Nonconforming Cell Product | 1 | 1
Completed | 37 | 81
Not Completed | 55 | 11
Not completed — Adverse Event | 1 | 0
Not completed — Death | 2 | 2
Not completed — Death due to the COVID-19 pandemic | 0 | 1
Not completed — Lack of Efficacy | 28 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 3 | 0
Not completed — Disease relapse | 15 | 6
Not completed — Study drug manufacturing failure | 0 | 1
Not completed — other reasons | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Arm | Liso-cel Arm | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.2 (13.94) | 58.3 (12.61) | 56.3 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 48 | 79
  Male | 61 | 44 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 62 | 65 | 127
  Unknown or Not Reported | 27 | 24 | 51
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 10 | 18
  Black or African American | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 55 | 54 | 109
  Not Collected or Reported | 25 | 22 | 47
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) Per Independent Review Committee (IRC)
Description: Time from randomization to death, progressive disease (PD), failure to achieve complete response (CR) or partial response (PR) by 9 weeks or start of new antineoplastic therapy, whichever occurs first. CR: Target nodes masses must regress to ≤ 1.5cm in LDi, no extralymphatic sites, no new lesions. PR: ≥ 50% decrease in sum of diameters of up to 6 target nodes and extranodal sites, no new lesions, spleen must have regressed > 50% in length. PD: LDi > 1.5cm, increase by ≥ 50% from PPD nadir, an increase in LDi or SDi from nadir, 0.5 cm for lesions ≤ 2cm, 1.0cm for lesions > 2cm. Complete metabolic response: Lymph nodes score 1, 2, 3 with/without residual mass on 5-point scale, no new lesions, no FDG-avid disease. Partial metabolic response: Lymph nodes score 4 or 5, reduced uptake from baseline, no new lesions, residual uptake higher than normal, reduced from baseline. Progressive metabolic disease: Score 4 or 5 with an increase in uptake intensity from baseline and/or new FDG-avid.
Time Frame: From randomization to death from any cause, PD, failure to achieve CR or PR by 9 weeks post randomization, or start of new antineoplastic therapy due to efficacy concerns, whichever occurs first (Up to 36 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Standard of Care Arm: 3 cycles of standard of care (SOC) salvage therapy (R-DHAP, R-ICE and R-GDP) per physician's choice. Participants responding to SOC are expected to undergo high dose chemotherapy (HDCT) and hematopoietic stem cell transplant (HSCT). If requested by the investigator, participants may be allowed to receive JCAR017 upon meeting progression, relapse, or suboptimal response. 1 cycle = 3 weeks
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 92 | 92
Months | 2.4 [2.2 to 4.9] | 29.5 [9.5 to NA] — Upper limit not calculated due to insufficient number of events per Kaplan-Meier product-limit estimates.

2. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete response rate (CRR) is defined as the percentage of participants achieving a best overall response of complete response (CR). Participants with unknown or missing response will be counted as non-evaluable in the analysis. CR: Target nodes/nodal masses must regress to ≤ 1.5 cm in LDi, no extralymphatic sites, no new lesions. Complete metabolic response: Lymph nodes/extralymphatic sites score 1, 2, 3 with/without residual mass on 5-point scale, no new lesions, no FDG-avid disease.
Time Frame: From randomization up to 3 years post randomization (Up to 36 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 92 | 92
Percentage of participants | 43.5 [33.2 to 54.2] | 73.9 [63.7 to 82.5]

3. Secondary Outcome: Number of Participants With Complete Response (CR)
Description: The number of participants achieving a best overall response of complete response (CR). Participants with unknown or missing response will be counted as non-evaluable in the analysis. CR: Target nodes/nodal masses must regress to ≤ 1.5 cm in LDi, no extralymphatic sites, no new lesions. Complete metabolic response: Lymph nodes/extralymphatic sites score 1, 2, 3 with/without residual mass on 5-point scale, no new lesions, no FDG-avid disease.
Time Frame: From randomization up to 3 years post randomization (Up to 36 months)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 92 | 92
Participants | 40 | 68

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from randomization to progressive disease (PD) or death from any cause, whichever occurs first. Estimates of time to event are from Kaplan-Meier product-limit estimates. PD: LDi > 1.5 cm, increase by ≥ 50% from PPD nadir, an increase in LDi or SDi from nadir, 0.5 cm for lesions ≤ 2 cm, 1.0 cm for lesions > 2 cm. Progressive metabolic disease: Score 4 or 5 with an increase in the intensity of uptake from baseline and/or new FDG-avid.
Time Frame: From randomization to progression, or death from any cause, whichever occurs first (Up to 36 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 92 | 92
Months | 6.2 [4.3 to 8.6] | NA [12.6 to NA] — Median and upper limit not calculated due to insufficient number of events per Kaplan-Meier product-limit estimates.

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from randomization to death due to any cause. Estimates of time to event are from Kaplan-Meier product-limit estimates.
Time Frame: From randomization to time of death due to any cause (Up to 36 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 92 | 92
Months | NA [18.2 to NA] — Median and upper limit not calculated due to insufficient number of events per Kaplan-Meier product-limit estimates. | NA [42.8 to NA] — Median and upper limit not calculated due to insufficient number of events per Kaplan-Meier product-limit estimates.

6. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants achieving a best overall response of partial response (PR) or complete response (CR). CR: Target nodes masses must regress to ≤ 1.5cm in LDi, no extralymphatic sites, no new lesions. PR: ≥ 50% decrease in sum of diameters of up to 6 target nodes and extranodal sites, no new lesions, spleen must have regressed > 50% in length. Complete metabolic response: Lymph nodes score 1, 2, 3 with/without residual mass on 5-point scale, no new lesions, no FDG-avid disease. Partial metabolic response: Lymph nodes score 4 or 5, reduced uptake from baseline, no new lesions, residual uptake higher than normal, reduced from baseline.
Time Frame: From randomization to PR or CR (Up to 36 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 92 | 92
Percentage of participants | 48.9 [38.3 to 59.6] | 87.0 [78.3 to 93.1]

7. Secondary Outcome: Duration of Response (DoR) Per Independent Review Committee (IRC)
Description: DoR is defined as the time from first partial or complete response (CR or PR) to disease progression, start of new antineoplastic therapy due to efficacy concerns or death, whichever occurs first. CR: Target nodes masses must regress to ≤ 1.5cm in LDi, no extralymphatic sites, no new lesions. PR: ≥ 50% decrease in sum of diameters of up to 6 target nodes and extranodal sites, no new lesions, spleen must have regressed > 50% in length. PD: LDi > 1.5cm, increase by ≥ 50% from PPD nadir, an increase in LDi or SDi from nadir, 0.5 cm for lesions ≤ 2cm, 1.0cm for lesions > 2cm. Complete metabolic response: Lymph nodes score 1, 2, 3 with/without residual mass on 5-point scale, no new lesions, no FDG-avid disease. Partial metabolic response: Lymph nodes score 4 or 5, reduced uptake from baseline, no new lesions, residual uptake higher than normal, reduced from baseline. Progressive metabolic disease: Score 4 or 5 with an increase in uptake intensity from baseline and/or new FDG-avid.
Time Frame: From randomization to to disease progression, start of new antineoplastic therapy due to efficacy concerns or death, whichever occurs first (Up to 36 months)
Population: All randomized participants with PR or CR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 45 | 80
Months | 9.1 [5.1 to NA] — Upper limit not calculated due to insufficient number of events per Kaplan-Meier product-limit estimates. | NA [16.9 to NA] — Median and upper limit not calculated due to insufficient number of events per Kaplan-Meier product-limit estimates.

8. Secondary Outcome: Number of Participants With Progression-free Survival on Next Line of Treatment (PFS-2)
Description: Progression-free Survival (PFS)-2 based on investigator's assessment is defined as time from randomization to second objective progressive disease (PD) or death from any cause, whichever occurs first. Estimates of time to event are from Kaplan-Meier product-limit estimates. PD: LDi > 1.5 cm, increase by ≥ 50% from PPD nadir, an increase in LDi or SDi from nadir, 0.5 cm for lesions ≤ 2 cm, 1.0 cm for lesions > 2 cm. Progressive metabolic disease: Score 4 or 5 with an increase in the intensity of uptake from baseline and/or new FDG-avid.
Time Frame: From randomization to second objective progression, or death from any cause, whichever occurs first (Up to 36 months)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 92 | 92
Participants
  Number of patients who died | 15 | 10
  Number of patients with first progression | 60 | 40
  Number of patients with second progression | 8 | 8

9. Secondary Outcome: Event-free Survival (EFS) Rate
Description: EFS rate is defined as the percentage of participants free of any EFS event at fixed timepoints. Complete response: Target nodes masses must regress to ≤ 1.5cm in LDi, no extralymphatic sites, no new lesions. Partial response: ≥ 50% decrease in sum of diameters of up to 6 target nodes and extranodal sites, no new lesions, spleen must have regressed > 50% in length. Progression: LDi > 1.5cm, increase by ≥ 50% from PPD nadir, an increase in LDi or SDi from nadir, 0.5 cm for lesions ≤ 2cm, 1.0cm for lesions > 2cm. Complete metabolic response: Lymph nodes score 1, 2, 3 with/without residual mass on 5-point scale, no new lesions, no FDG-avid disease. Partial metabolic response: Lymph nodes score 4 or 5, reduced uptake from baseline, no new lesions, residual uptake higher than normal, reduced from baseline. Metabolic progression: Score 4 or 5 with an increase in uptake intensity from baseline and/or new FDG-avid.
Time Frame: Months 6, 12, 18, 24, 36
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 92 | 92
Percentage of participants
  EFS Rate at 6 months | 36.2 [26.3 to 46.1] | 68.1 [58.6 to 77.7]
  EFS Rate at 12 months | 22.6 [13.9 to 31.3] | 57.0 [46.8 to 67.2]
  EFS Rate at 18 months | 22.6 [13.9 to 31.3] | 52.6 [42.3 to 62.8]
  EFS Rate at 24 months | 21.5 [13.0 to 30.0] | 51.4 [41.1 to 61.7]
  EFS Rate at 36 months | 19.1 [11.0 to 27.3] | 45.8 [35.2 to 56.5]

10. Secondary Outcome: Progression-free Survival (PFS) Rate
Description: Progression-free Survival (PFS) rate is defined as the percentage of participants free of any PFS event at fixed timepoints. Progression-free survival is defined as the time from randomization to progressive disease (PD) or death from any cause, whichever occurs first. Estimates of time to event are from Kaplan-Meier product-limit estimates. PD: LDi > 1.5 cm, increase by ≥ 50% from PPD nadir, an increase in LDi or SDi from nadir, 0.5 cm for lesions ≤ 2 cm, 1.0 cm for lesions > 2 cm. Progressive metabolic disease: Score 4 or 5 with an increase in the intensity of uptake from baseline and/or new FDG-avid.
Time Frame: Months 6, 12, 18, 24, 36
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 92 | 92
Percentage of participants
  PFS Rate at 6 months | 51.7 [40.2 to 63.1] | 73.7 [64.5 to 83.0]
  PFS Rate at 12 months | 31.3 [20.3 to 42.4] | 63.0 [52.8 to 73.2]
  PFS Rate at 18 months | 31.3 [20.3 to 42.4] | 58.2 [47.7 to 68.7]
  PFS Rate at 24 months | 29.7 [18.8 to 40.7] | 57.0 [46.4 to 67.5]
  PFS Rate at 36 months | 26.5 [15.9 to 37.1] | 50.9 [39.9 to 62.0]

11. Secondary Outcome: Overall Survival (OS) Rate
Description: Overall Survival (OS) rate is defined as the percentage of participants alive at fixed timepoints. OS is defined as the time from randomization to death due to any cause. Participants alive or lost to follow up at the time of analysis will be censored at the last date the participants was known to be alive.
Time Frame: Months 6, 12, 18, 24, 36
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 92 | 92
Percentage of participants
  OS Rate at 6 months | 88.9 [82.4 to 95.4] | 93.4 [88.4 to 98.5]
  OS Rate at 12 months | 72.0 [62.7 to 81.3] | 83.5 [75.8 to 91.1]
  OS Rate at 18 months | 61.7 [51.5 to 71.8] | 73.3 [64.2 to 82.5]
  OS Rate at 24 months | 58.2 [47.9 to 68.5] | 67.5 [57.8 to 77.2]
  OS Rate at 36 months | 51.8 [41.2 to 62.4] | 62.8 [52.7 to 72.9]
  Participants who died | 45.7 [NA to NA] — Only percentage of participants who died to be reported | 37.0 [NA to NA] — Only percentage of participants who died to be reported
  Participants who were censored | 54.3 [NA to NA] — Only percentage of participants who were censored to be reported | 63.0 [NA to NA] — Only percentage of participants who were censored to be reported

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment that does not necessarily have a causal relation with this treatment. TEAEs are adverse events occurring or worsening on or after the date of randomization and within 90 days after last dose of chemotherapy (Arm A), or within 90 days after the infusion of JCAR017 (Arm B) or start of new antineoplastic therapy, whichever occurs first as well as those AEs made known to the investigator at any time thereafter that are suspected of being related to study treatment. Graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From randomization to 90 days after last dose or start of new antineoplastic therapy, whichever occurs first (Up to 16.5 months)
Population: All participants treated in any study medication per overall participants and in clinical, histological and molecular subgroups that are prespecified for this endpoint (subgroups are not mutually exclusive)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 91 | 92
Participants
  Overall participants with TEAEs | 90 | 92
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL) with TEAEs: number analyzed (Participants) | 58 | 60
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL) with TEAEs | 57 | 60
  NIH: Follicular Lymphoma Grade 3B with TEAEs: number analyzed (Participants) | 0 | 1
  NIH: Follicular Lymphoma Grade 3B with TEAEs |  | 1
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology with TEAEs: number analyzed (Participants) | 20 | 22
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology with TEAEs | 20 | 22
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma with TEAEs: number analyzed (Participants) | 9 | 8
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma with TEAEs | 9 | 8
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma with TEAEs: number analyzed (Participants) | 4 | 1
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma with TEAEs | 4 | 1
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo with TEAEs: number analyzed (Participants) | 50 | 53
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo with TEAEs | 49 | 53
  DLBCL: DLBCL from Transformed Indolent NHL with TEAEs: number analyzed (Participants) | 8 | 7
  DLBCL: DLBCL from Transformed Indolent NHL with TEAEs | 8 | 7

13. Secondary Outcome: Number of Participants With Serious Treatment-Emergent Adverse Events (TEAEs)
Description: A serious adverse event is defined as any adverse event occurring at any dose that results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or constitutes an important medical event. Treatment emergent adverse events are adverse events occurring or worsening on or after the date of randomization and within 90 days after last dose of chemotherapy (Arm A), or within 90 days after the infusion of JCAR017 (Arm B) or start of new antineoplastic therapy, whichever occurs first as well as those AEs made known to the investigator at any time thereafter that are suspected of being related to study treatment. Graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 91 | 92
Participants
  Overall Participants with serious TEAEs | 45 | 43
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL) with serious TEAEs: number analyzed (Participants) | 58 | 60
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL) with serious TEAEs | 29 | 23
  NIH: Follicular Lymphoma Grade 3B with serious TEAEs: number analyzed (Participants) | 0 | 1
  NIH: Follicular Lymphoma Grade 3B with serious TEAEs |  | 0
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology with serious TEAEs: number analyzed (Participants) | 20 | 22
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology with serious TEAEs | 9 | 17
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma with serious TEAEs: number analyzed (Participants) | 9 | 8
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma with serious TEAEs | 4 | 2
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma with serious TEAEs: number analyzed (Participants) | 4 | 1
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma with serious TEAEs | 3 | 1
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo with serious TEAEs: number analyzed (Participants) | 50 | 53
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo with serious TEAEs | 25 | 20
  DLBCL: DLBCL from Transformed Indolent NHL with serious TEAEs: number analyzed (Participants) | 8 | 7
  DLBCL: DLBCL from Transformed Indolent NHL with serious TEAEs | 4 | 3

14. Secondary Outcome: Change From Baseline in Hematology Parameters 1: Hemoglobin
Description: Change from baseline in hemoglobin. Baseline value will be defined as the last value on the randomization date (+3 days) or before the date/time of randomization (date if date/time not collected).
Time Frame: baseline, months 1, 2, 3, 4, 6, 9, 12, 18, 24, 36
Population: All treated participants with a baseline value and a post-baseline value at the time point
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 73 | 84
g/L
  Hemoglobin Month 1 | -16.98 (13.408) | -14.94 (14.628)
  Hemoglobin Month 2: number analyzed (Participants) | 1 | 0
  Hemoglobin Month 2 | -25.00 (NA) — insufficient number of participants to calculate standard deviation |
  Hemoglobin Month 3: number analyzed (Participants) | 41 | 72
  Hemoglobin Month 3 | -30.83 (19.013) | -15.78 (19.410)
  Hemoglobin Month 4: number analyzed (Participants) | 1 | 0
  Hemoglobin Month 4 | -22.00 (NA) — insufficient number of participants to calculate standard deviation |
  Hemoglobin Month 6: number analyzed (Participants) | 30 | 62
  Hemoglobin Month 6 | -6.80 (14.935) | -3.16 (19.755)
  Hemoglobin Month 9: number analyzed (Participants) | 22 | 60
  Hemoglobin Month 9 | 0.36 (19.242) | -0.52 (15.632)
  Hemoglobin Month 12: number analyzed (Participants) | 18 | 59
  Hemoglobin Month 12 | 6.17 (14.598) | 3.32 (15.417)
  Hemoglobin Month 18: number analyzed (Participants) | 19 | 52
  Hemoglobin Month 18 | 11.37 (14.592) | 7.38 (12.854)
  Hemoglobin Month 24: number analyzed (Participants) | 17 | 45
  Hemoglobin Month 24 | 13.88 (18.996) | 7.38 (16.986)
  Hemoglobin Month 36: number analyzed (Participants) | 17 | 41
  Hemoglobin Month 36 | 14.41 (16.978) | 13.63 (12.417)

15. Secondary Outcome: Change From Baseline in Selected Hematology Parameters 2
Description: Change from baseline in selected hematology parameters such as leukocytes, lymphocytes, neutrophils, and platelets. Baseline value will be defined as the last value on the randomization date (+3 days) or before the date/time of randomization (date if date/time not collected).
Time Frame: baseline, months 1, 2, 3, 4, 6, 9, 12, 18, 24, 36
Population: All treated participants with a baseline value and a post-baseline value at the time point
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 73 | 84
10^9 cells/L
  Month 1 leukocytes | 0.815 (6.9413) | -3.219 (2.4688)
  Month 2 leukocytes: number analyzed (Participants) | 1 | 0
  Month 2 leukocytes | -0.870 (NA) — insufficient number of participants to calculate standard deviation |
  Month 3 leukocytes: number analyzed (Participants) | 41 | 72
  Month 3 leukocytes | -3.445 (5.8845) | -2.234 (2.3520)
  Month 4 leukocytes: number analyzed (Participants) | 1 | 0
  Month 4 leukocytes | -1.180 (NA) — insufficient number of participants to calculate standard deviation |
  Month 6 leukocytes: number analyzed (Participants) | 30 | 62
  Month 6 leukocytes | -1.699 (1.9099) | -1.853 (2.5876)
  Month 9 leukocytes: number analyzed (Participants) | 22 | 60
  Month 9 leukocytes | -0.710 (3.0670) | -1.156 (3.3604)
  Month 12 leukocytes: number analyzed (Participants) | 18 | 59
  Month 12 leukocytes | -0.427 (1.4093) | -1.138 (2.3772)
  Month 18 leukocytes: number analyzed (Participants) | 19 | 52
  Month 18 leukocytes | -0.598 (1.6136) | -1.088 (2.8028)
  Month 24 leukocytes: number analyzed (Participants) | 17 | 45
  Month 24 leukocytes | 0.694 (3.0465) | -0.806 (2.5709)
  Month 36 leukocytes: number analyzed (Participants) | 17 | 41
  Month 36 leukocytes | 0.761 (2.3637) | -0.970 (3.0158)
  Month 1 lymphocytes: number analyzed (Participants) | 73 | 83
  Month 1 lymphocytes | -0.2824 (0.43519) | -0.7380 (0.43499)
  Month 2 lymphocytes: number analyzed (Participants) | 1 | 0
  Month 2 lymphocytes | -0.2100 (NA) — insufficient number of participants to calculate standard deviation |
  Month 3 lymphocytes: number analyzed (Participants) | 19 | 71
  Month 3 lymphocytes | -0.4216 (0.55872) | -0.1318 (0.43385)
  Month 4 lymphocytes: number analyzed (Participants) | 1 | 0
  Month 4 lymphocytes | -0.1700 (NA) — insufficient number of participants to calculate standard deviation |
  Month 6 lymphocytes: number analyzed (Participants) | 30 | 62
  Month 6 lymphocytes | 0.1343 (0.38219) | -0.0845 (0.48047)
  Month 9 lymphocytes: number analyzed (Participants) | 22 | 60
  Month 9 lymphocytes | 0.3264 (0.66121) | -0.0442 (0.39684)
  Month 12 lymphocytes: number analyzed (Participants) | 18 | 59
  Month 12 lymphocytes | 0.5089 (0.71831) | 0.0097 (0.37252)
  Month 18 lymphocytes: number analyzed (Participants) | 19 | 52
  Month 18 lymphocytes | 0.6942 (0.98993) | 0.2283 (0.55421)
  Month 24 lymphocytes: number analyzed (Participants) | 17 | 45
  Month 24 lymphocytes | 0.8688 (1.12695) | 0.3298 (0.51386)
  Month 36 lymphocytes: number analyzed (Participants) | 17 | 40
  Month 36 lymphocytes | 1.2253 (1.20268) | 0.3550 (0.55387)
  Month 1 neutrophils: number analyzed (Participants) | 73 | 83
  Month 1 neutrophils | 1.368 (6.5393) | -2.065 (2.3479)
  Month 2 neutrophils: number analyzed (Participants) | 1 | 0
  Month 2 neutrophils | -0.590 (NA) — insufficient number of participants to calculate standard deviation |
  Month 3 neutrophils: number analyzed (Participants) | 19 | 71
  Month 3 neutrophils | -0.621 (6.8377) | -1.909 (2.1727)
  Month 4 neutrophils: number analyzed (Participants) | 1 | 0
  Month 4 neutrophils | -1.160 (NA) — insufficient number of participants to calculate standard deviation |
  Month 6 neutrophils: number analyzed (Participants) | 30 | 62
  Month 6 neutrophils | -1.648 (1.7635) | -1.584 (2.4539)
  Month 9 neutrophils: number analyzed (Participants) | 22 | 60
  Month 9 neutrophils | -0.879 (2.9777) | -1.001 (3.1318)
  Month 12 neutrophils: number analyzed (Participants) | 18 | 59
  Month 12 neutrophils | -0.822 (1.5780) | -1.035 (2.2898)
  Month 18 neutrophils: number analyzed (Participants) | 19 | 52
  Month 18 neutrophils | -1.167 (1.3772) | -1.189 (2.6342)
  Month 24 neutrophils: number analyzed (Participants) | 17 | 45
  Month 24 neutrophils | -0.124 (2.5434) | -0.998 (2.5506)
  Month 36 neutrophils: number analyzed (Participants) | 17 | 40
  Month 36 neutrophils | -0.404 (1.8392) | -0.998 (2.5222)
  Month 1 platelets: number analyzed (Participants) | 72 | 78
  Month 1 platelets | 13.9 (140.94) | 29.4 (115.53)
  Month 2 platelets: number analyzed (Participants) | 1 | 0
  Month 2 platelets | 13.0 (NA) — insufficient number of participants to calculate standard deviation |
  Month 3 platelets: number analyzed (Participants) | 38 | 71
  Month 3 platelets | -189.5 (132.93) | -65.7 (100.52)
  Month 4 platelets: number analyzed (Participants) | 1 | 0
  Month 4 platelets | -74.0 (NA) — insufficient number of participants to calculate standard deviation |
  Month 6 platelets: number analyzed (Participants) | 30 | 60
  Month 6 platelets | -45.5 (94.13) | -48.2 (89.04)
  Month 9 platelets: number analyzed (Participants) | 22 | 58
  Month 9 platelets | -57.0 (110.48) | -48.9 (89.29)
  Month 12 platelets: number analyzed (Participants) | 18 | 56
  Month 12 platelets | -66.5 (85.82) | -42.4 (92.65)
  Month 18 platelets: number analyzed (Participants) | 19 | 52
  Month 18 platelets | -68.0 (84.69) | -32.6 (81.68)
  Month 24 platelets: number analyzed (Participants) | 17 | 44
  Month 24 platelets | -29.4 (103.87) | -28.7 (79.70)
  Month 36 platelets: number analyzed (Participants) | 17 | 40
  Month 36 platelets | -45.2 (123.28) | -10.5 (72.79)

16. Secondary Outcome: Change From Baseline in Selected Chemistry Parameters 1
Description: Change from baseline in selected chemistry parameters such as alanine aminotransferase, aspartate aminotransferase, and lactate dehydrogenase. Baseline value will be defined as the last value on the randomization date (+3 days) or before the date/time of randomization (date if date/time not collected).
Time Frame: baseline, months 1, 2, 3, 4, 6, 9, 12, 18, 24, 36
Population: All treated participants with a baseline value and a post-baseline value at the time point
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 76 | 88
U/L
  Month 1 Alanine Aminotransferase | 17.22 (25.997) | -0.52 (18.337)
  Month 2 Alanine Aminotransferase: number analyzed (Participants) | 1 | 0
  Month 2 Alanine Aminotransferase | 4.00 (NA) — insufficient number of participants to calculate standard deviation |
  Month 3 Alanine Aminotransferase: number analyzed (Participants) | 43 | 73
  Month 3 Alanine Aminotransferase | -3.40 (22.295) | 2.53 (13.246)
  Month 4 Alanine Aminotransferase: number analyzed (Participants) | 1 | 0
  Month 4 Alanine Aminotransferase | -3.00 (NA) — insufficient number of participants to calculate standard deviation |
  Month 6 Alanine Aminotransferase: number analyzed (Participants) | 31 | 65
  Month 6 Alanine Aminotransferase | 2.81 (21.067) | 3.08 (14.813)
  Month 9 Alanine Aminotransferase: number analyzed (Participants) | 23 | 61
  Month 9 Alanine Aminotransferase | 2.43 (20.165) | 5.23 (16.660)
  Month 12 Alanine Aminotransferase: number analyzed (Participants) | 18 | 58
  Month 12 Alanine Aminotransferase | 0.72 (23.542) | 4.19 (19.653)
  Month 18 Alanine Aminotransferase: number analyzed (Participants) | 20 | 53
  Month 18 Alanine Aminotransferase | 10.40 (15.892) | -0.45 (10.943)
  Month 24 Alanine Aminotransferase: number analyzed (Participants) | 16 | 48
  Month 24 Alanine Aminotransferase | 7.69 (15.134) | 1.88 (13.211)
  Month 36 Alanine Aminotransferase: number analyzed (Participants) | 17 | 41
  Month 36 Alanine Aminotransferase | 12.41 (17.429) | 13.98 (104.054)
  Month 1 Aspartate Aminotransferase: number analyzed (Participants) | 75 | 87
  Month 1 Aspartate Aminotransferase | 3.38 (16.624) | 2.03 (17.526)
  Month 2 Aspartate Aminotransferase: number analyzed (Participants) | 1 | 0
  Month 2 Aspartate Aminotransferase | 5.00 (NA) — insufficient number of participants to calculate standard deviation |
  Month 3 Aspartate Aminotransferase: number analyzed (Participants) | 43 | 71
  Month 3 Aspartate Aminotransferase | -6.47 (17.248) | -1.24 (8.800)
  Month 4 Aspartate Aminotransferase: number analyzed (Participants) | 1 | 0
  Month 4 Aspartate Aminotransferase | 3.00 (NA) — insufficient number of participants to calculate standard deviation |
  Month 6 Aspartate Aminotransferase: number analyzed (Participants) | 30 | 65
  Month 6 Aspartate Aminotransferase | 1.23 (15.911) | 1.78 (8.550)
  Month 9 Aspartate Aminotransferase: number analyzed (Participants) | 22 | 60
  Month 9 Aspartate Aminotransferase | 3.68 (12.549) | 2.12 (10.355)
  Month 12 Aspartate Aminotransferase: number analyzed (Participants) | 18 | 57
  Month 12 Aspartate Aminotransferase | -1.44 (16.180) | 1.88 (13.200)
  Month 18 Aspartate Aminotransferase: number analyzed (Participants) | 20 | 54
  Month 18 Aspartate Aminotransferase | 4.90 (7.663) | -1.22 (7.452)
  Month 24 Aspartate Aminotransferase: number analyzed (Participants) | 16 | 48
  Month 24 Aspartate Aminotransferase | 4.63 (9.172) | 0.90 (10.757)
  Month 36 Aspartate Aminotransferase: number analyzed (Participants) | 18 | 40
  Month 36 Aspartate Aminotransferase | 9.06 (15.117) | 14.95 (94.651)
  Month 1 Lactate Dehydrogenase: number analyzed (Participants) | 70 | 73
  Month 1 Lactate Dehydrogenase | -66.7 (222.79) | -14.0 (203.18)
  Month 2 Lactate Dehydrogenase: number analyzed (Participants) | 1 | 0
  Month 2 Lactate Dehydrogenase | 27.0 (NA) — insufficient number of participants to calculate standard deviation |
  Month 3 Lactate Dehydrogenase: number analyzed (Participants) | 40 | 64
  Month 3 Lactate Dehydrogenase | -57.2 (377.22) | -84.1 (183.29)
  Month 4 Lactate Dehydrogenase: number analyzed (Participants) | 1 | 0
  Month 4 Lactate Dehydrogenase | 117.0 (NA) — insufficient number of participants to calculate standard deviation |
  Month 6 Lactate Dehydrogenase: number analyzed (Participants) | 25 | 56
  Month 6 Lactate Dehydrogenase | -85.5 (310.71) | -53.7 (183.53)
  Month 9 Lactate Dehydrogenase: number analyzed (Participants) | 20 | 50
  Month 9 Lactate Dehydrogenase | -85.0 (362.52) | -62.0 (186.25)
  Month 12 Lactate Dehydrogenase: number analyzed (Participants) | 18 | 48
  Month 12 Lactate Dehydrogenase | -52.9 (74.56) | -41.9 (207.30)
  Month 18 Lactate Dehydrogenase: number analyzed (Participants) | 17 | 43
  Month 18 Lactate Dehydrogenase | -44.1 (71.19) | -50.8 (133.31)
  Month 24 Lactate Dehydrogenase: number analyzed (Participants) | 15 | 38
  Month 24 Lactate Dehydrogenase | -45.6 (75.04) | -63.3 (148.25)
  Month 36 Lactate Dehydrogenase: number analyzed (Participants) | 12 | 31
  Month 36 Lactate Dehydrogenase | -46.0 (85.14) | -59.9 (124.62)

17. Secondary Outcome: Change From Baseline in Selected Chemistry Parameters 2
Description: Change from baseline in selected chemistry parameters such as magnesium, phosphate, potassium, and sodium. Baseline value will be defined as the last value on the randomization date (+3 days) or before the date/time of randomization (date if date/time not collected).
Time Frame: baseline, months 1, 2, 3, 4, 6, 9, 12, 18, 24, 36
Population: All treated participants with a baseline value and a post-baseline value at the time point
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 76 | 88
mmol/L
  Month 1 magnesium | -0.023 (0.1145) | 0.009 (0.0933)
  Month 2 magnesium: number analyzed (Participants) | 1 | 0
  Month 2 magnesium | -0.080 (NA) — insufficient number of participants to calculate standard deviation |
  Month 3 magnesium: number analyzed (Participants) | 44 | 73
  Month 3 magnesium | -0.063 (0.1210) | 0.007 (0.1010)
  Month 4 magnesium: number analyzed (Participants) | 1 | 0
  Month 4 magnesium | -0.200 (NA) — insufficient number of participants to calculate standard deviation |
  Month 6 magnesium: number analyzed (Participants) | 31 | 66
  Month 6 magnesium | -0.041 (0.1452) | 0.015 (0.1090)
  Month 9 magnesium: number analyzed (Participants) | 23 | 62
  Month 9 magnesium | -0.027 (0.1459) | 0.025 (0.1079)
  Month 12 magnesium: number analyzed (Participants) | 18 | 58
  Month 12 magnesium | 0.012 (0.1047) | 0.031 (0.1054)
  Month 18 magnesium: number analyzed (Participants) | 20 | 54
  Month 18 magnesium | 0.033 (0.0639) | 0.032 (0.1065)
  Month 24 magnesium: number analyzed (Participants) | 16 | 48
  Month 24 magnesium | 0.040 (0.1145) | 0.015 (0.1027)
  Month 36 magnesium: number analyzed (Participants) | 18 | 41
  Month 36 magnesium | 0.039 (0.0920) | 0.011 (0.0751)
  Month 1 phosphate | -0.061 (0.2643) | -0.038 (0.2498)
  Month 2 phosphate: number analyzed (Participants) | 1 | 0
  Month 2 phosphate | 0.030 (NA) — insufficient number of participants to calculate standard deviation |
  Month 3 phosphate: number analyzed (Participants) | 44 | 74
  Month 3 phosphate | -0.128 (0.3299) | 0.039 (0.2316)
  Month 4 phosphate: number analyzed (Participants) | 1 | 0
  Month 4 phosphate | 0.130 (NA) — insufficient number of participants to calculate standard deviation |
  Month 6 phosphate: number analyzed (Participants) | 31 | 66
  Month 6 phosphate | 0.140 (0.2166) | -0.020 (0.2276)
  Month 9 phosphate: number analyzed (Participants) | 23 | 62
  Month 9 phosphate | 0.025 (0.2020) | -0.028 (0.2098)
  Month 12 phosphate: number analyzed (Participants) | 18 | 59
  Month 12 phosphate | -0.021 (0.1578) | -0.090 (0.2051)
  Month 18 phosphate: number analyzed (Participants) | 20 | 54
  Month 18 phosphate | -0.025 (0.2666) | -0.059 (0.2224)
  Month 24 phosphate: number analyzed (Participants) | 16 | 48
  Month 24 phosphate | -0.064 (0.2469) | -0.061 (0.2549)
  Month 36 phosphate: number analyzed (Participants) | 18 | 41
  Month 36 phosphate | -0.044 (0.2464) | -0.061 (0.2053)
  Month 1 potassium: number analyzed (Participants) | 75 | 88
  Month 1 potassium | -0.08 (0.400) | -0.05 (0.460)
  Month 2 potassium: number analyzed (Participants) | 1 | 0
  Month 2 potassium | 0.30 (NA) — insufficient number of participants to calculate standard deviation |
  Month 3 potassium: number analyzed (Participants) | 43 | 73
  Month 3 potassium | -0.33 (0.604) | 0.00 (0.428)
  Month 4 potassium: number analyzed (Participants) | 1 | 0
  Month 4 potassium | 0.80 (NA) — insufficient number of participants to calculate standard deviation |
  Month 6 potassium: number analyzed (Participants) | 31 | 66
  Month 6 potassium | 0.11 (0.337) | 0.08 (0.359)
  Month 9 potassium: number analyzed (Participants) | 23 | 62
  Month 9 potassium | -0.06 (0.447) | 0.12 (0.391)
  Month 12 potassium: number analyzed (Participants) | 18 | 58
  Month 12 potassium | 0.01 (0.445) | 0.06 (0.491)
  Month 18 potassium: number analyzed (Participants) | 20 | 54
  Month 18 potassium | 0.06 (0.380) | 0.15 (0.411)
  Month 24 potassium: number analyzed (Participants) | 16 | 48
  Month 24 potassium | 0.09 (0.516) | 0.09 (0.435)
  Month 36 potassium: number analyzed (Participants) | 18 | 40
  Month 36 potassium | 0.07 (0.549) | 0.11 (0.430)
  month 1 sodium: number analyzed (Participants) | 75 | 88
  month 1 sodium | -2.75 (3.493) | -1.09 (2.875)
  month 2 sodium: number analyzed (Participants) | 1 | 0
  month 2 sodium | -1.00 (NA) — insufficient number of participants to calculate standard deviation |
  month 3 sodium: number analyzed (Participants) | 44 | 73
  month 3 sodium | -1.86 (4.496) | 0.59 (3.054)
  month 4 sodium: number analyzed (Participants) | 1 | 0
  month 4 sodium | -2.00 (NA) — insufficient number of participants to calculate standard deviation |
  month 6 sodium: number analyzed (Participants) | 31 | 66
  month 6 sodium | -0.42 (2.514) | 0.33 (3.222)
  month 9 sodium: number analyzed (Participants) | 23 | 61
  month 9 sodium | 0.52 (2.108) | -0.08 (3.111)
  month 12 sodium: number analyzed (Participants) | 18 | 58
  month 12 sodium | 0.33 (2.114) | -0.34 (4.046)
  month 18 sodium: number analyzed (Participants) | 20 | 54
  month 18 sodium | 0.45 (2.964) | 0.74 (3.572)
  month 24 sodium: number analyzed (Participants) | 16 | 48
  month 24 sodium | -1.00 (3.246) | 1.02 (3.795)
  month 36 sodium: number analyzed (Participants) | 18 | 40
  month 36 sodium | -0.44 (2.229) | 0.25 (3.432)

18. Secondary Outcome: Overall Response Rate (ORR) by Subgroups
Description: as for outcome 6
Time Frame: From randomization to PR or CR (Up to 36 months)
Population: All randomized participants per clinical, histological and molecular subgroups that are pre-specified for ORR (subgroups are not mutually exclusive and participants are not exclusive to one subgroup)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 72 | 70
Percentage of participants
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL): number analyzed (Participants) | 58 | 60
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL) | 51.7 [38.2 to 65.0] | 86.7 [75.4 to 94.1]
  NIH: Follicular Lymphoma Grade 3B: number analyzed (Participants) | 0 | 1
  NIH: Follicular Lymphoma Grade 3B |  | 100 [2.5 to 100.0]
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology: number analyzed (Participants) | 21 | 22
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology | 42.9 [21.8 to 66.0] | 81.8 [59.7 to 94.8]
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma: number analyzed (Participants) | 9 | 8
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma | 33.3 [7.5 to 70.1] | 100 [63.1 to 100.0]
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma: number analyzed (Participants) | 4 | 1
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma | 75.0 [19.4 to 99.4] | 100 [2.5 to 100.0]
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo: number analyzed (Participants) | 50 | 53
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo | 54.0 [39.3 to 68.2] | 86.8 [74.7 to 94.5]
  DLBCL: DLBCL from Transformed Indolent NHL: number analyzed (Participants) | 8 | 7
  DLBCL: DLBCL from Transformed Indolent NHL | 37.5 [8.5 to 75.5] | 85.7 [42.1 to 99.6]
  DLBCL: Germinal Center B-cell like (GCB): number analyzed (Participants) | 40 | 45
  DLBCL: Germinal Center B-cell like (GCB) | 50.0 [33.8 to 66.2] | 91.1 [78.8 to 97.5]
  DLBCL: Activated B-cell-like, non-GCB: number analyzed (Participants) | 29 | 21
  DLBCL: Activated B-cell-like, non-GCB | 44.8 [26.4 to 64.3] | 85.7 [63.7 to 97.0]
  NHL: Double-hit lymphoma (DBL)/triple-hit lymphoma (THL): number analyzed (Participants) | 20 | 22
  NHL: Double-hit lymphoma (DBL)/triple-hit lymphoma (THL) | 40.0 [19.1 to 63.9] | 81.8 [59.7 to 94.8]
  NHL: Non-DHL/THL | 51.4 [39.3 to 63.3] | 88.6 [78.7 to 94.9]

19. Secondary Outcome: Event-free Survival (EFS) by Subgroups
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All randomized participants per clinical, histological and molecular subgroups that are pre-specified for EFS (subgroups are not mutually exclusive)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 72 | 70
Months
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL): number analyzed (Participants) | 58 | 60
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL) | 3.0 [2.2 to 6.4] | NA [9.5 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NIH: Follicular Lymphoma Grade 3B: number analyzed (Participants) | 0 | 1
  NIH: Follicular Lymphoma Grade 3B |  | NA [NA to NA] — Median, the lower bound and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology: number analyzed (Participants) | 21 | 22
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology | 2.2 [0.9 to 3.9] | 4.6 [4.1 to 12.6]
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma: number analyzed (Participants) | 9 | 8
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma | 2.2 [1.0 to NA] — The upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [11.0 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma: number analyzed (Participants) | 4 | 1
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma | NA [2.3 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [NA to NA] — Median, the lower bound and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo: number analyzed (Participants) | 50 | 53
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo | 4.4 [2.2 to 7.5] | 33.2 [9.4 to NA] — The upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  DLBCL: DLBCL from Transformed Indolent NHL: number analyzed (Participants) | 8 | 7
  DLBCL: DLBCL from Transformed Indolent NHL | 2.1 [1.2 to 11.2] | NA [1.9 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  DLBCL: Germinal Center B-cell like (GCB): number analyzed (Participants) | 40 | 45
  DLBCL: Germinal Center B-cell like (GCB) | 2.1 [1.6 to 4.9] | 11.7 [6.0 to NA] — The upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  DLBCL: Activated B-cell-like, non-GCB: number analyzed (Participants) | 29 | 21
  DLBCL: Activated B-cell-like, non-GCB | 2.3 [2.1 to 7.5] | 33.2 [4.9 to NA] — The upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NHL: Double-hit lymphoma (DBL)/triple-hit lymphoma (THL): number analyzed (Participants) | 20 | 22
  NHL: Double-hit lymphoma (DBL)/triple-hit lymphoma (THL) | 2.1 [0.9 to 3.9] | 4.6 [4.1 to 12.6]
  NHL: Non-DHL/THL | 2.8 [2.2 to 6.4] | NA [15.6 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events

20. Secondary Outcome: Progression-free Survival (PFS) by Subgroups
Description: as for outcome 4
Time Frame: From randomization to progression, or death from any cause, whichever occurs first (Up to 36 months)
Population: All randomized participants per clinical, histological and molecular subgroups that are pre-specified for PFS (subgroups are not mutually exclusive)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 72 | 70
Months
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL): number analyzed (Participants) | 58 | 60
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL) | 6.0 [2.9 to 8.6] | NA [30.9 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NIH: Follicular Lymphoma Grade 3B: number analyzed (Participants) | 0 | 1
  NIH: Follicular Lymphoma Grade 3B |  | NA [NA to NA] — Median, the lower bound and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology: number analyzed (Participants) | 21 | 22
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology | 4.3 [1.4 to 6.5] | 5.8 [4.3 to 14.8]
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma: number analyzed (Participants) | 9 | 8
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma | NA [1.0 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [11.0 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma: number analyzed (Participants) | 4 | 1
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma | NA [28.2 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [NA to NA] — Median, the lower bound and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo: number analyzed (Participants) | 50 | 53
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo | 6.4 [3.1 to 8.6] | NA [12.2 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  DLBCL: DLBCL from Transformed Indolent NHL: number analyzed (Participants) | 8 | 7
  DLBCL: DLBCL from Transformed Indolent NHL | 3.4 [1.2 to NA] — the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [2.3 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  DLBCL: Germinal Center B-cell like (GCB): number analyzed (Participants) | 40 | 45
  DLBCL: Germinal Center B-cell like (GCB) | 4.6 [2.0 to 6.4] | 14.8 [6.2 to NA] — the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  DLBCL: Activated B-cell-like, non-GCB: number analyzed (Participants) | 29 | 21
  DLBCL: Activated B-cell-like, non-GCB | 7.5 [2.3 to 9.4] | 33.2 [6.6 to NA] — the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NHL: Double-hit lymphoma (DBL)/triple-hit lymphoma (THL): number analyzed (Participants) | 20 | 22
  NHL: Double-hit lymphoma (DBL)/triple-hit lymphoma (THL) | 4.3 [1.4 to 6.5] | 5.8 [4.3 to 14.8]
  NHL: Non-DHL/THL | 6.4 [4.6 to 9.4] | NA [33.2 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events

21. Secondary Outcome: Overall Survival (OS) by Subgroups
Description: as for outcome 5
Time Frame: From randomization to time of death due to any cause (Up to 36 months)
Population: All randomized participants per clinical, histological and molecular subgroups that are pre-specified for OS (subgroups are not mutually exclusive)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 72 | 70
Months
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL): number analyzed (Participants) | 58 | 60
  Non-Hodgkin Lymphoma (NHL): Diffuse Large B-cell Lymphoma (DLBCL) | NA [17.0 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [42.8 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NIH: Follicular Lymphoma Grade 3B: number analyzed (Participants) | 0 | 1
  NIH: Follicular Lymphoma Grade 3B |  | NA [NA to NA] — Median, the lower bound and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology: number analyzed (Participants) | 21 | 22
  NIH: High-Grade B-cell Lymphoma with DLBCL Histology | 16.3 [5.3 to NA] — The upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | 13.3 [7.9 to NA] — The upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma: number analyzed (Participants) | 9 | 8
  NIH: Primary Mediastinal (thymic) Large B-cell Lymphoma | NA [17.9 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [11.0 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma: number analyzed (Participants) | 4 | 1
  NIH: T Cell/Histiocyte-Rich Large B-Cell Lymphoma | NA [8.9 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [NA to NA] — Median, the lower bound and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo: number analyzed (Participants) | 50 | 53
  Diffuse Large B-cell Lymphoma (DLBCL): DLBCL NOS de novo | NA [16.7 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [42.8 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  DLBCL: DLBCL from Transformed Indolent NHL: number analyzed (Participants) | 8 | 7
  DLBCL: DLBCL from Transformed Indolent NHL | 28.2 [2.0 to NA] — The upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [14.2 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  DLBCL: Germinal Center B-cell like (GCB): number analyzed (Participants) | 40 | 45
  DLBCL: Germinal Center B-cell like (GCB) | NA [18.2 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [15.8 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  DLBCL: Activated B-cell-like, non-GCB: number analyzed (Participants) | 29 | 21
  DLBCL: Activated B-cell-like, non-GCB | 16.3 [9.7 to NA] — The upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [32.4 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NHL: Double-hit lymphoma (DBL)/triple-hit lymphoma (THL): number analyzed (Participants) | 20 | 22
  NHL: Double-hit lymphoma (DBL)/triple-hit lymphoma (THL) | 16.3 [5.3 to 30.7] | 13.3 [7.9 to NA] — The upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events
  NHL: Non-DHL/THL | NA [27.5 to NA] — Median and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events | NA [NA to NA] — Median, the lower bound and the upper bound of the 95% Confidence Interval could not be calculated due to insufficient number of participants with events

22. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer - Quality of Life C30 Questionnaire (EORTC QLQ-C30)
Description: Change from baseline in EORTC QLQ-C30 specified parameters including global health/quality of life, cognitive functioning, physical functioning, and fatigue. It is composed of both multi-item scales and single item measures. All of the scales and single-item measures range in score from 0 to 100. A 10-point change in the scoring is considered to be a meaningful change in HRQoL. Functional scale and global health status/HRQoL higher scale score represents a higher level of well-being and better ability of daily functioning. Symptom scale/item higher score represents a high level of symptomatic problem. Baseline value will be defined as the last value on the randomization date (+3 days) or before the date/time of randomization (date if date/time not collected).
Time Frame: baseline, months 1, 6, 9, 12, 18, 24, 36
Population: All treated participants with a health-related quality of life baseline assessment value and a post-baseline value at the time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 41 | 43
score on a scale
  Global Health/Quality of Life Month 1 | -9.55 (25.655) | -5.23 (18.004)
  Global Health/Quality of Life Month 6: number analyzed (Participants) | 15 | 29
  Global Health/Quality of Life Month 6 | -2.78 (24.734) | 12.36 (23.635)
  Global Health/Quality of Life Month 9: number analyzed (Participants) | 11 | 24
  Global Health/Quality of Life Month 9 | 5.30 (24.516) | 12.50 (22.252)
  Global Health/Quality of Life Month 12: number analyzed (Participants) | 8 | 28
  Global Health/Quality of Life Month 12 | 15.63 (32.865) | 8.93 (24.525)
  Global Health/Quality of Life Month 18: number analyzed (Participants) | 9 | 24
  Global Health/Quality of Life Month 18 | 14.81 (29.397) | 8.33 (23.442)
  Global Health/Quality of Life Month 24: number analyzed (Participants) | 10 | 24
  Global Health/Quality of Life Month 24 | 12.50 (28.934) | 7.29 (23.093)
  Global Health/Quality of Life Month 36: number analyzed (Participants) | 10 | 25
  Global Health/Quality of Life Month 36 | 15.00 (21.802) | 2.67 (21.071)
  Physical Functioning Month 1 | -8.94 (19.867) | -4.03 (16.339)
  Physical Functioning Month 6: number analyzed (Participants) | 16 | 29
  Physical Functioning Month 6 | -2.08 (11.081) | 2.24 (17.470)
  Physical Functioning Month 9: number analyzed (Participants) | 11 | 24
  Physical Functioning Month 9 | 0.61 (9.167) | 5.00 (21.825)
  Physical Functioning Month 12: number analyzed (Participants) | 8 | 28
  Physical Functioning Month 12 | 10.00 (17.817) | 4.52 (17.875)
  Physical Functioning Month 18: number analyzed (Participants) | 9 | 25
  Physical Functioning Month 18 | 13.33 (22.608) | 1.73 (17.027)
  Physical Functioning Month 24: number analyzed (Participants) | 10 | 24
  Physical Functioning Month 24 | 10.67 (18.645) | 2.78 (22.147)
  Physical Functioning Month 36: number analyzed (Participants) | 10 | 25
  Physical Functioning Month 36 | 7.33 (15.540) | -1.87 (16.613)
  Cognitive Functioning Month 1 | -8.54 (19.047) | -0.39 (16.462)
  Cognitive Functioning Month 6: number analyzed (Participants) | 15 | 29
  Cognitive Functioning Month 6 | -3.33 (14.365) | 3.45 (20.596)
  Cognitive Functioning Month 9: number analyzed (Participants) | 11 | 24
  Cognitive Functioning Month 9 | -3.03 (16.361) | 9.72 (23.008)
  Cognitive Functioning Month 12: number analyzed (Participants) | 8 | 28
  Cognitive Functioning Month 12 | -4.17 (7.715) | 4.17 (27.074)
  Cognitive Functioning Month 18: number analyzed (Participants) | 9 | 24
  Cognitive Functioning Month 18 | 0.00 (18.634) | 4.17 (26.580)
  Cognitive Functioning Month 24: number analyzed (Participants) | 10 | 24
  Cognitive Functioning Month 24 | 0.00 (13.608) | 0.00 (26.919)
  Cognitive Functioning Month 36: number analyzed (Participants) | 10 | 25
  Cognitive Functioning Month 36 | -1.67 (9.461) | 2.67 (17.795)
  Fatigue Month 1 | 19.24 (24.848) | 0.26 (20.501)
  Fatigue Month 6: number analyzed (Participants) | 16 | 29
  Fatigue Month 6 | 0.69 (27.657) | -12.84 (29.811)
  Fatigue Month 9: number analyzed (Participants) | 11 | 24
  Fatigue Month 9 | -4.04 (29.090) | -10.65 (36.702)
  Fatigue Month 12: number analyzed (Participants) | 8 | 28
  Fatigue Month 12 | -6.94 (8.267) | -9.52 (33.363)
  Fatigue Month 18: number analyzed (Participants) | 9 | 25
  Fatigue Month 18 | -6.17 (22.299) | -10.22 (30.919)
  Fatigue Month 24: number analyzed (Participants) | 10 | 24
  Fatigue Month 24 | -6.67 (19.030) | -8.80 (30.557)
  Fatigue Month 36: number analyzed (Participants) | 10 | 25
  Fatigue Month 36 | -3.33 (16.605) | -5.33 (25.884)

23. Secondary Outcome: Change From Baseline in the Functional Assessment of Cancer Therapy-Lymphoma Subscale (FACT-Lym)
Description: Change from Baseline in the Functional Assessment of Cancer Therapy-Lymphoma 15-item lymphoma-specific "Additional concerns" subscale (FACT-Lym). The LYM items are scored on a 0 ("Not at all") to 4 ("Very much") response scale. Items are aggregated to a single score on a 0-60 scale. Baseline value will be defined as the last value on the randomization date (+3 days) or before the date/time of randomization (date if date/time not collected). A meaningful change from baseline in the FACT-Lym score, often referred to as the minimally important difference (MID), typically ranges between 6.5 and 11.2 points for the total score. This range indicates a clinically significant improvement or deterioration in a patient's health-related quality of life.
Time Frame: baseline, months 1, 6, 9, 12, 18, 24, 36
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 38 | 40
score on a scale
  Month 1 | -0.76 (5.558) | 0.35 (7.329)
  Month 6: number analyzed (Participants) | 16 | 29
  Month 6 | 2.19 (9.474) | 3.52 (10.805)
  Month 9: number analyzed (Participants) | 9 | 23
  Month 9 | 0.11 (9.597) | 5.48 (14.330)
  Month 12: number analyzed (Participants) | 7 | 27
  Month 12 | 5.43 (3.645) | 3.93 (13.485)
  Month 18: number analyzed (Participants) | 8 | 25
  Month 18 | 3.50 (5.632) | 2.56 (12.149)
  Month 24: number analyzed (Participants) | 10 | 22
  Month 24 | 5.20 (5.789) | 2.18 (12.374)
  Month 36: number analyzed (Participants) | 10 | 24
  Month 36 | 4.90 (5.152) | 0.50 (9.478)

24. Secondary Outcome: Hospital Resource Utilization (HRU) Results
Description: Hospital resource utilization (HRU) results including hospitalized, reasons for hospitalizations, and admitted to intensive care unit (ICU)
Time Frame: Up to 36 months
Population: All participants treated in any study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 91 | 92
Participants
  Hospitalized | 74 | 87
  Hospitalized due to Adverse Event (AE) | 42 | 44
  Hospitalized due to Progression of Disease | 2 | 6
  Hospitalized per protocol | 11 | 22
  Hospitalized due to other reasons | 56 | 71
  Admitted to Intensive Care Unit (ICU) | 4 | 5

25. Secondary Outcome: Percentage of Participants Completing High Dose Chemotherapy (HDCT)
Description: Percentage of Participants Completing High Dose Chemotherapy (HDCT).
Time Frame: Up to 5 months after first dose
Population: All treated participants in SOC arm
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 91 | 0
Percentage of participants | 47.3 |

26. Secondary Outcome: Percentage of Participants Completing Hematopoietic Stem Cell Transplant (HSCT)
Description: Percentage of Participants Completing Hematopoietic Stem Cell Transplant (HSCT).
Time Frame: Up to 5 months after first dose
Population: All treated participants in SOC arm
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care Arm | Liso-cel Arm
Number analyzed (Participants) | 91 | 0
Percentage of participants | 47.3 |

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from first dose until study completion (assessed up to approximately 60 months). SAEs and Other AEs were assessed from first dose to 90 days after last dose of study therapy (Up to 16.5 months).
Description: The number at Risk for All-Cause Mortality=All randomized participants. The number at Risk for SAEs and Other AEs=All treated participants.
  Randomized SOC (92) for All-Cause Mortality is presented separately under "SOC pre-crossover only" and "SOC-JCAR017 Pre- and post-cross over" arms as pre-specified
  Treated SOC (91) for SAEs and Other AEs is presented separately under "SOC pre-crossover only" and "SOC-JCAR017 Pre- and post-cross over" arms as pre-specified
Groups:
- SOC Arm (Pre-crossover Only): Participants received 3 cycles of standard of care (SOC) salvage therapy (R-DHAP, R-ICE and R-GDP) per physician's choice. Participants responding to SOC are expected to undergo high dose chemotherapy (HDCT) and hematopoietic stem cell transplant (HSCT). 1 cycle = 3 weeks
- Liso-cel Arm Only: [Lymphodepleting chemotherapy (LDC)] Fludarabine IV (30 mg/m^2/day for 3 days) and cyclophosphamide IV (300 mg/m^2/day for 3 days) followed by JCAR017 IV infusion at a dose of 100 x 10^6 JCAR017-positive viable transduced T cells (CAR+ T cells) on Day 29 (2 to 7 days after completion of LD chemotherapy)
- SOC-JCAR017 Arm Pre- and Post-Crossover (All Crossed): participants received 3 cycles of standard of care (SOC) salvage therapy (R-DHAP, R-ICE and R-GDP) per physician's choice. Participants responding to SOC are expected to undergo high dose chemotherapy (HDCT) and hematopoietic stem cell transplant (HSCT). Participants crossed over to JCAR017 regardless of if they received CAR T therapy or not.
Arm/Group | SOC Arm (Pre-crossover Only) | Liso-cel Arm Only | SOC-JCAR017 Arm Pre- and Post-Crossover (All Crossed)
All-Cause Mortality (participants affected / at risk) | 9/31 | 34/92 | 33/61
Serious Adverse Events (participants affected / at risk) | 21/30 | 43/92 | 19/61
Other Adverse Events (participants affected / at risk) | 30/30 | 92/92 | 57/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOC Arm (Pre-crossover Only) (N=30) | Liso-cel Arm Only (N=92) | SOC-JCAR017 Arm Pre- and Post-Crossover (All Crossed) (N=61)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Cytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 7 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 7 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 2 | 6 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 12 | 5
Engraftment syndrome (Immune system disorders) | 1 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Device related bacteraemia (Infections and infestations) | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0
Septic shock (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 2 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOC Arm (Pre-crossover Only) (N=30) | Liso-cel Arm Only (N=92) | SOC-JCAR017 Arm Pre- and Post-Crossover (All Crossed) (N=61)
Anaemia (Blood and lymphatic system disorders) | 20 | 62 | 24
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 10 | 1
Leukopenia (Blood and lymphatic system disorders) | 7 | 17 | 5
Lymphopenia (Blood and lymphatic system disorders) | 4 | 25 | 9
Neutropenia (Blood and lymphatic system disorders) | 14 | 75 | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 54 | 21
Sinus tachycardia (Cardiac disorders) | 2 | 7 | 2
Tachycardia (Cardiac disorders) | 5 | 9 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 6 | 2
Vision blurred (Eye disorders) | 1 | 6 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 13 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 30 | 10
Diarrhoea (Gastrointestinal disorders) | 14 | 23 | 9
Dry mouth (Gastrointestinal disorders) | 3 | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 5 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 1
Haematochezia (Gastrointestinal disorders) | 2 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 2 | 1
Nausea (Gastrointestinal disorders) | 17 | 49 | 14
Oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 3 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 6 | 1
Vomiting (Gastrointestinal disorders) | 10 | 18 | 6
Asthenia (General disorders) | 3 | 11 | 3
Chills (General disorders) | 0 | 8 | 4
Fatigue (General disorders) | 10 | 37 | 12
Mucosal inflammation (General disorders) | 5 | 5 | 0
Non-cardiac chest pain (General disorders) | 1 | 5 | 2
Oedema peripheral (General disorders) | 4 | 15 | 7
Pyrexia (General disorders) | 6 | 22 | 6
Cytokine release syndrome (Immune system disorders) | 0 | 33 | 24
Hypogammaglobulinaemia (Immune system disorders) | 0 | 9 | 2
COVID-19 (Infections and infestations) | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 2 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 6 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 4 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 8 | 1
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 6 | 0
Alanine aminotransferase increased (Investigations) | 3 | 6 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 6 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 8 | 4
Blood creatinine increased (Investigations) | 2 | 6 | 3
C-reactive protein increased (Investigations) | 2 | 1 | 1
International normalised ratio increased (Investigations) | 2 | 4 | 1
Neutrophil count decreased (Investigations) | 0 | 7 | 3
Platelet count decreased (Investigations) | 1 | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 12 | 21 | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 6 | 4
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 6 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 7 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 21 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 15 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 9 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 7 | 5
Malnutrition (Metabolism and nutrition disorders) | 4 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 17 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 14 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 12 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 11 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 7 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 8 | 4
Dizziness (Nervous system disorders) | 1 | 22 | 10
Dysgeusia (Nervous system disorders) | 3 | 3 | 0
Headache (Nervous system disorders) | 8 | 40 | 16
Paraesthesia (Nervous system disorders) | 2 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 7 | 2
Tremor (Nervous system disorders) | 0 | 11 | 10
Anxiety (Psychiatric disorders) | 1 | 5 | 1
Confusional state (Psychiatric disorders) | 0 | 5 | 6
Depression (Psychiatric disorders) | 2 | 4 | 2
Insomnia (Psychiatric disorders) | 5 | 19 | 4
Acute kidney injury (Renal and urinary disorders) | 2 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 13 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 13 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 7 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 9 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 3 | 8 | 4
Hypotension (Vascular disorders) | 2 | 19 | 10
Jugular vein thrombosis (Vascular disorders) | 2 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT03575351/Prot_SAP_000.pdf